CLINICAL TRIAL: NCT02218853
Title: Psychosis and Affective Research Domains and Intermediate Phenotypes
Acronym: PARDIP
Status: Completed | Type: Observational
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: Beth Israel Deaconess Medical Center (Other); Hartford Hospital (Other); University of Georgia (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Other Study IDs: MH077851; 1R01MH096913-01A1 (NIH)
Record Dates: First submitted 2014-08-11; First posted 2014-08-18 (Estimated); Last update posted 2019-09-19 (Actual); Status verified 2019-09

CONDITIONS: Bipolar I Disorder, Unspecified, With Psychotic Features; Bipolar I Disorder, Unspecified, Without Psychotic Features
Keywords: Bipolar disorder; Psychosis; Schizophrenia
MeSH Terms: conditions — Bipolar Disorder; Psychotic Disorders; Schizophrenia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA will be extracted from blood (or buccal swab) and stored at the UT Southwestern Human Genetic Center in a departmental freezer at -80 degrees. Part of the blood sample will be used to create an immortalized lymphocyte culture (a lymphoblastoid cell line) for future genetic analysis, and will be stored in a Cell Bank at the UT Southwestern Human Genetic Center. The blood samples will be labeled by a coded identifier (number) and will not be personally identifiable. Only specifically designated research staff from Dr. Tamminga's group and from the UT Southwestern Human Genetic Center will have an access to stored DNA samples. All samples will be de-identified. The genetic data will be in password-protected computers in the Investigators' research offices.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Bipolar I disorder, with psychosis: Individuals diagnosed with Bipolar I disorder, with psychotic features
- Bipolar I disorder, without psychosis: Individuals diagnosed with Bipolar I disorder, without psychotic features
- Healthy Controls: Must have no personal history of any psychotic or mood disorder, or a family history of psychotic or recurrent mood disorder among their first-degree relatives

SUMMARY:
The objective of this multi-site research collaboration is to test the manifestation and distribution of biological markers for psychosis and affect dimensions across the schizophrenia/bipolar (SZ-BD) diagnostic boundary, and to examine heritability and genetic associations for these biological markers.

DETAILED DESCRIPTION:
The B-SNIP research consortium previously obtained dense phenotypes across the psychosis spectrum in an effort to observe features both (i) distinctive to and (ii) shared between DSM-type categorical diagnoses. Despite the broad range of extra-clinical phenotypes, we had limited success finding clinical SZ-BD diagnosis-specific features; instead, most phenotypes were distributed continuously across DSM diagnoses. To describe more biologically homogeneous groups, therefore, we combined all psychosis probands and implemented a multi-stage analysis procedure, beginning with identification of psychosis biomarkers (variables with the largest effect sizes for differentiating psychosis and healthy groups) including cognitive, electrophysiological, and oculo-motor measures ('classical' endophenotypes). We then estimated the number of subgroups that efficiently optimized variance among the biomarkers (n=3) and differentiated the individual psychosis cases into these subgroups. Subsequently, the subgroups were tested for biological uniqueness using meaningful external validators (structural and functional brain imaging, social functioning, and familial data). Given the neurobiological distinctiveness of these subgroups, we called them psychosis Biotypes. DSM diagnoses were distributed across all Biotypes. Compared to DSM diagnoses, Biotype membership enhanced group separations on biomarkers. These results indicate that groups of psychosis cases can be generated with homogeneous phenotypic characteristics independent of DSM diagnoses. The proposed study aims to further develop Biotype definitions and demonstrate that psychosis Biotypes constructed from a dense biomarker panel (i) are replicable, (ii) neurobiologically distinctive, and (iii) have unique genetic characteristics.

ELIGIBILITY:
Inclusion Criteria:

* Must provide consent to participate after being fully informed about the study procedures and the information to be collected
* Males and females
* Ages 18-60 years old
* All races and ethnicities
* Probands: Must meet DSM-IV criteria for bipolar I disorder with or without lifetime history of psychosis; Healthy Controls: Must have no personal history of any psychotic or mood disorder, or a family history of psychotic or recurrent mood disorder among their first-degree relatives
* Must be judged to be capable of completing the study procedures by study investigators
* Must be able to read, speak, and understand English

Exclusion Criteria:

* An estimated IQ<70
* Major neurological or cognitive disorder (e.g., seizure disorder, traumatic brain injury, cerebrovascular disease, pervasive developmental disorder)
* Serious medical, neuro-ophthalmological, or neurological illness that could affect CNS functioning (e.g., decompensated cardiovascular disease, decompensated chronic obstructive pulmonary disease, late stages of diabetes, AIDS)
* DSM-IV diagnosis of alcohol or illicit substance abuse within 1 month, or alcohol or substance dependence within 3 months, or extensive history of past substance use
* Women who are pregnant (due to unknown risks related to MRI exposure)
* Presence of medical (e.g., artificial joints, brain aneurism clips, surgical pins, rods, wires, implants) or non-medical (e.g., metal piercing) irremovable metallic objects on/inside body (due to MRI-relevant risks)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study population will be comprised of individuals between the ages of 18-60 years old who meet DSM-IV criteria for Bipolar I disorder, read/speak/understand the English language, and are deemed capable of completing the study procedures by the research investigators.
Sampling Method: Probability Sample
Enrollment: 113 (Actual)
Dates: Start 2014-04; Primary Completion 2017-06 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Differences in those with Bipolar disorder with psychosis, without psychosis, and healthy controls on functional and structural brain imaging, neurocognitive assessments, and neurophysiological tests | One day

SECONDARY OUTCOMES:
Differences in those with Bipolar disorder with psychosis, without psychosis, and healthy controls on clinical assessment questionnaires | One day
  The investigators will assess clustering of probands and relatives across composite biomarkers independent of diagnostic status using multivariate taxometric procedures.

OTHER OUTCOMES:
Differences in those with Bipolar disorder with psychosis, without psychosis, and healthy controls in DNA and dermal biopsy sampling | One day
  The investigators will collect DNA from all proband and relative subjects and collaboratively sequence the genetic material to associate genes with specific biomarkers and composite Biotype definitions. We will also collect plasma and cellular specimens to bank for analysis of additional molecular biomarkers unique to each Biotype.

CONTACTS AND LOCATIONS:
Overall Officials: Carol A Tamminga, M.D., Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States

REFERENCES:
- See also: Tamminga Lab and Clinic Website — http://www.utsouthwestern.edu/labs/schizophrenia/